CLINICAL TRIAL: NCT00597727
Title: A Double-blinded, Placebo-controlled Study of Peanut Sublingual Immunotherapy in Children - DBPC Peanut SLIT
Brief Title: A Study of Sublingual Immunotherapy in Peanut-allergic Children
Acronym: SLB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-2296; 5R01AT004435-09 (NIH)
Record Dates: First submitted 2008-01-07; First posted 2008-01-18 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2017-04

CONDITIONS: Food Hypersensitivity
Keywords: Peanut Allergy; Sublingual immunotherapy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: For the initial 12 months of the study, subjects were blinded to receive either peanut SLIT or placebo. After unblinding, subjects on placebo are crossed over to receive open-label peanut SLIT. They underwent an identical dosing protocol as those that were initially randomized to active treatment.
  After 12 months of peanut SLIT dosing, whether initially randomized to active or crossed over from placebo, all subjects remained part of an open-label extended maintenance phase for the duration of the study (total peanut SLIT dosing 36-60 months)
  2 additional cohorts were included in the protocol. One cohort, called the Early Unblinded Peanut SLIT cohort, was unblinded prior to the scheduled 12 month time point for pharmacy safety concerns. The second cohort, called the Pilot Peanut SLIT Rollover cohort involved subjects from the prior pilot study (NCT00429429) who were added to the study through an amendment and received open-label peanut SLIT.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Blinded Peanut SLIT (Active Comparator): Blinded subjects who received peanut sublingual drops for the initial 12 month blinded phase of the study.
  Interventions: Drug: Peanut SLIT
- Blinded Placebo SLIT (Placebo Comparator): Blinded subjects who received placebo sublingual drops for the initial 12 month blinded phase of the study.
  Interventions: Drug: Placebo SLIT
- Ext. maint. open label peanut SLIT (Other): After completing the blinded phase of the study, subjects receiving Blinded Peanut SLIT continued on extended maintenance open-label peanut SLIT for the duration of the study. Subjects receiving Blinded Placebo SLIT were crossed over and underwent the 12 month buildup protocol on open label peanut SLIT and then continued on extended maintenance treatment for the duration of the study.
  Interventions: Drug: Peanut SLIT
- Early unblinded peanut SLIT (Other): Subjects who were unblinded prematurely during the blinded phase of the study and then re-enrolled as an open label cohort.
  Interventions: Drug: Peanut SLIT
- Pilot peanut SLIT rollover cohort (Other): Subjects from the original phase 1 study of peanut SLIT (NCT00429429) who were rolled over into the current protocol as an open label peanut SLIT cohort.
  Interventions: Drug: Peanut SLIT

INTERVENTIONS:
Drug: Peanut SLIT — Liquid peanut protein drops diluted in glycerin which are dosed under the tongue.
  Other Names: Sublingual peanut protein drops
  Arms: Blinded Peanut SLIT; Early unblinded peanut SLIT; Ext. maint. open label peanut SLIT; Pilot peanut SLIT rollover cohort
Drug: Placebo SLIT — Liquid glycerin without peanut which are dosed under the tongue.
  Other Names: Sublingual glycerin saline drops
  Arms: Blinded Placebo SLIT

SUMMARY:
The specific aim of this study is to determine if peanut allergen-specific SLIT will cause clinical desensitization and tolerance to develop in peanut-allergic young children.

DETAILED DESCRIPTION:
In spite of increased recognition and understanding of food allergies, food-induced anaphylaxis remains the single most common cause of anaphylaxis seen in hospital emergency departments, accounting for about one third of anaphylaxis cases seen. It is estimated that about 30,000 food-induced anaphylactic events are seen in U.S. emergency departments each year and that about 200 fatal cases occur in the U.S. each year. Either peanuts or tree nuts cause more than 80% of these reactions. No treatments are available and avoidance is the only approved intervention.

The goal of this study is to investigate peanut sublingual immunotherapy (SLIT) as a treatment for children with peanut allergy. This study is primarily designed to evaluate the efficacy and safety of peanut SLIT compared to placebo after 12 months. Secondarily, the study is designed to evaluate the efficacy of extended maintenance dosing of peanut SLIT in inducing lasting tolerance after discontinuation of the peanut SLIT. Mechanistic studies will be completed concurrently as exploratory endpoints to understand changes in the allergic immune response related to peanut SLIT.

ELIGIBILITY:
Inclusion Criteria:

* Peanut IgE > 7kU/L (> 2kU/L for children aged 2 years and under) AND
* History of significant clinical symptoms within 60 minutes after the ingestion of peanuts.

Exclusion Criteria:

* History of severe life-threatening anaphylaxis to peanut, OR
* Medical history that would prevent a DBPCFC to peanut, OR
* Subjects with wheat or oat allergy (which are used in the placebo), OR
* Unable to cooperate with challenge procedures, OR
* Unable to be reached by telephone for follow-up

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin SJ, Vickery BP, Kulis MD, Kim EH, Varshney P, Steele P, Kamilaris J, Hiegel AM, Carlisle SK, Smith PB, Scurlock AM, Jones SM, Burks AW. Sublingual versus oral immunotherapy for peanut-allergic children: a retrospective comparison. J Allergy Clin Immunol. 2013 Aug;132(2):476-8.e2. doi: 10.1016/j.jaci.2013.02.017. Epub 2013 Mar 25. No abstract available. PMID 23534975
- [Result] Kim EH, Bird JA, Kulis M, Laubach S, Pons L, Shreffler W, Steele P, Kamilaris J, Vickery B, Burks AW. Sublingual immunotherapy for peanut allergy: clinical and immunologic evidence of desensitization. J Allergy Clin Immunol. 2011 Mar;127(3):640-6.e1. doi: 10.1016/j.jaci.2010.12.1083. Epub 2011 Feb 1. PMID 21281959
- [Result] Kulis M, Saba K, Kim EH, Bird JA, Kamilaris N, Vickery BP, Staats H, Burks AW. Increased peanut-specific IgA levels in saliva correlate with food challenge outcomes after peanut sublingual immunotherapy. J Allergy Clin Immunol. 2012 Apr;129(4):1159-62. doi: 10.1016/j.jaci.2011.11.045. Epub 2012 Jan 10. PMID 22236732

RESULTS

PARTICIPANT FLOW:
Groups:
- Ext Maint Open Label Peanut SLIT: After completing the blinded phase of the study, subjects receiving Blinded Peanut SLIT continued on extended maintenance open-label peanut SLIT for the duration of the study. Subjects receiving Blinded Placebo SLIT were crossed over and underwent the 12 month buildup protocol on open label peanut SLIT and then continued on extended maintenance treatment for the duration of the study.
Period: 12 Month Blinded Phase
Arm/Group | Blinded Peanut SLIT | Blinded Placebo SLIT | Ext Maint Open Label Peanut SLIT | Early Unblinded Peanut SLIT | Pilot Peanut SLIT Rollover Cohort
Started | 14 | 15 | 0 | 27 | 4
Completed | 14 | 15 | 0 | 17 | 3
Not Completed | 0 | 0 | 0 | 10 | 1
Period: Open-label Extended Maintenance Phase
Arm/Group | Blinded Peanut SLIT | Blinded Placebo SLIT | Ext Maint Open Label Peanut SLIT | Early Unblinded Peanut SLIT | Pilot Peanut SLIT Rollover Cohort
Started | 0 (Blinded peanut SLIT + blinded placebo SLIT continued in Ext Open Label Peanut SLIT after unblinding) | 0 (Blinded peanut SLIT + blinded placebo SLIT continued in Ext Open Label Peanut SLIT after unblinding) | 29 (Blinded peanut SLIT + blinded placebo SLIT continued in Ext Open Label Peanut SLIT after unblinding.) | 17 | 3
Completed | 0 | 0 | 23 | 14 | 1
Not Completed | 0 | 0 | 6 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Blinded Peanut SLIT: Blinded subjects who received peanut sublingual drops) at the beginning of the study.
- Blinded Placebo SLIT: Blinded subjects who receive placebo (glycerin sublingual drops) at the beginning of the study.
  Placebo SLIT: Liquid glycerin without peanut which are dosed under the tongue.
- Total: Total of all reporting groups
Arm/Group | Blinded Peanut SLIT | Blinded Placebo SLIT | Early Unblinded Peanut SLIT | Pilot Peanut SLIT Rollover Cohort | Total
Number analyzed (Participants) | 14 | 15 | 27 | 4 | 60
Age, Continuous [Median (Full Range); unit: years] | 6.0 [2.8 to 10.9] | 6.6 [1.6 to 11.9] | 6.0 [1.5 to 11.8] | 15.6 [8.9 to 20.8] | 6.4 [1.6 to 20.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 6 | 0 | 18
  Male | 9 | 8 | 21 | 4 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 15 | 27 | 4 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 13 | 14 | 24 | 3 | 54
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 27 | 4 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Can Tolerate the Peanut Oral Food Challenge After 12 Months of Peanut SLIT Dosing
Description: Upon completion of 12 months of peanut SLIT treatment, subjects underwent a double-blind placebo controlled food challenge (DBPCFC) to assess desensitization (an increase in reaction threshold while on therapy). A DBPCFC involves the ingestion of small increasing amounts of peanut up to a cumulative total amount. The primary clinical efficacy outcome of the study was the percentage of peanut allergic subjects who completed a 2500 mg peanut protein DBPCFC without developing symptoms after 12 months of peanut SLIT therapy.
Time Frame: 12 months
Population: Interim analysis in 7/2010 showed statistically significant difference in peanut tolerated during oral food challenge (OFC) by active treatment vs placebo (1710mg vs 85mg). Further OFCs for those on placebo was considered more risk than benefit thus were discontinued resulting in subsequent patients being unblinded after 12 months without an OFC
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Peanut SLIT | Blinded Placebo SLIT | Early Unblinded Peanut SLIT | Pilot Peanut SLIT Rollover Cohort
Number analyzed (Participants) | 11 | 7 | 17 | 3
percentage of participants | 45.5 | 0 | 11.8 | 66.7

2. Secondary Outcome: Percentage of Subjects Tolerating a Peanut Oral Food Challenge 2-4 Weeks After Discontining Peanut SLIT Dosing
Description: Upon completion of 36-60 months of peanut SLIT treatment, subjects underwent a double-blind placebo controlled food challenge (DBPCFC) to assess desensitization (an increase in reaction threshold while on therapy). A DBPCFC involves the ingestion of small increasing amounts of peanut up to a cumulative total amount. Peanut SLIT therapy was then discontinued for 2-4 weeks to assess for persistence of the desensitization response called sustained unresponsiveness (SU). The secondary clinical efficacy outcome of the study was the percentage of peanut allergic subjects who completed a 5000 mg peanut protein DBPCFC without developing symptoms 2-4 weeks after discontinuing peanut SLIT therapy.
Time Frame: 36-60 months
Population: Although the 12 month OFC was discontinued beginning in 7/2010, all subjects reaching the end of study (36-60 months of treatment) underwent an OFC resulting in more patients performing the end of study OFC than the 12 month OFC.
Measure: Number; unit: percentage of participants
Arm/Group | Ext Maint Open Label Peanut SLIT | Early Unblinded Peanut SLIT | Pilot Peanut SLIT Rollover Cohort
Number analyzed (Participants) | 23 | 14 | 1
percentage of participants | 26.1 | 28.6 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from the initial day of study drug dosing through unblinding after 12 months of therapy continuing through the extended maintenance phase for a total of 36-60 months of treatment concluding with the end of study DBPCFC 2-4 weeks off of peanut SLIT therapy.
Arm/Group | Blinded Peanut SLIT | Blinded Placebo SLIT | Ext Maint Open Label Peanut SLIT | Early Unblinded Peanut SLIT | Pilot Peanut SLIT Rollover Cohort
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/29 | 0/27 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/29 | 0/27 | 0/4
Other Adverse Events (participants affected / at risk) | 10/14 | 12/15 | 21/29 | 19/27 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Peanut SLIT (N=14) | Blinded Placebo SLIT (N=15) | Ext Maint Open Label Peanut SLIT (N=29) | Early Unblinded Peanut SLIT (N=27) | Pilot Peanut SLIT Rollover Cohort (N=4)
Vomiting (Gastrointestinal disorders) | 2 | 2 | 3 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0
Erythematous rash (Skin and subcutaneous tissue disorders) | 4 | 4 | 4 | 5 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0
Oropharyngeal itching (Skin and subcutaneous tissue disorders) | 8 | 7 | 17 | 13 | 1
Sneezing (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 2 | 0
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 7 | 2 | 0
Itchy nose (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 0
Skin itch (Skin and subcutaneous tissue disorders) | 3 | 6 | 8 | 3 | 0
Lip or eye swelling (Skin and subcutaneous tissue disorders) | 3 | 1 | 7 | 5 | 1
Eye itch (Eye disorders) | 0 | 1 | 4 | 1 | 0
Eye tearing (Eye disorders) | 1 | 1 | 1 | 2 | 0
Hives (Skin and subcutaneous tissue disorders) | 5 | 2 | 5 | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 6 | 1 | 19 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0

LIMITATIONS AND CAVEATS:
The initial 27 subjects in the study were unblinded in 12/2009 due to concerns for study drug integrity. These subjects were offered reentry into the study on open label drug. 18 accepted and are presented as the Early Unblinded Peanut SLIT cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No